CLINICAL TRIAL: NCT05120466
Title: Pilot Trial of a Novel Media Literacy Tobacco Prevention Program for High School Students
Brief Title: Media Literacy for High School Tobacco Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jaime Sidani, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY21020198
Record Dates: First submitted 2021-10-26; First posted 2021-11-15 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Adolescent Behavior; Tobacco Use; E-Cig Use
MeSH Terms: conditions — Adolescent Behavior; Tobacco Use; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Health Education Curriculum (Active Comparator): Students will receive the school's usual health education curriculum.
  Interventions: Behavioral: Usual health education curriculum
- Usual Health Education Curriculum plus Intervention (Experimental): Students will receive the school's usual health education curriculum. Students will also receive the intervention. Delivery of the intervention (i.e., timing, frequency) will be determined by discussing the results of the Aim 1 focus groups with teachers and administrators.
  Interventions: Behavioral: AD IT UP media literacy intervention; Behavioral: Usual health education curriculum

INTERVENTIONS:
Behavioral: AD IT UP media literacy intervention — AD IT UP was originally developed in 2006 as a classroom-based cigarette prevention program focused on traditional media influences, and was converted to a web-based program in 2011. In 2019, the AD IT UP program was updated substantially to include other forms of tobacco, such as e-cigarettes, and other forms of media, such as social media.
  Arms: Usual Health Education Curriculum plus Intervention
Behavioral: Usual health education curriculum — The school's regular health education curriculum includes classroom lectures, hands on activities and group work.

SUMMARY:
This research project will explore the feasibility and acceptability of a web-based media literacy tobacco prevention program. The project will be conducted with 9th or 10th graders in two high schools in Pittsburgh, Pennsylvania.

DETAILED DESCRIPTION:
Specific Aim 1: To assess students' preferences for delivery of the web-based media literacy tobacco prevention program. Investigators will conduct focus groups with students. Students will be shown clips from the program and asked to provide feedback about the preferred frequency and setting for the program.

Specific Aim 2: Investigators will conduct a pilot trial of the intervention via a cluster randomized controlled trial. The control group will receive their usual health education curriculum. The intervention group will receive their usual health education curriculum with the addition of the intervention. All students will be asked to complete a pre-test, a post-test, and two follow-up surveys (approximately 4 and 12 months post-intervention). Feasibility endpoints will include overall program completion, recruitment/attendance rates, and retention rates. Acceptability outcomes will assess student perceptions toward the intervention. A sub-aim will be to conduct focus groups and interviews with students, teachers, and administrators to assess implementation barriers and facilitators.

ELIGIBILITY:
Inclusion Criteria:

* 9th or 10th grade student
* enrolled at participating Pittsburgh-area school

Exclusion Criteria:

* Inability to read the surveys

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible 9th or 10th grade students recruited to participate in the study | 1 month
  Parents will be asked to return an opt out form if they do not want their student to participate. Students will provide assent if they wish to participate. Recruitment will be determined by calculating the percentage of eligible 9th or 10th grade students not opted out by their parents that also provide assent.
Percentage of participants retained through the final data collection | 12 months
  Retention will be calculated as the percentage of 9th or 10th grade students who completed the baseline survey and also completed the 12 month follow-up survey.
Percentage of participants indicating moderate to high acceptability of the AD IT UP program | post-test immediately following completion of the intervention
  Acceptability of the intervention will be assessed with closed-ended and open-ended items on the post-test survey immediately following completion of the intervention.
  Students will be asked on a 5-point Likert scale with responses ranging from Strongly Agree to Strongly Disagree (with a neutral middle) their agreement about the following: "I enjoyed AD IT UP," "I understood AD IT UP," "AD IT UP was easy to use," "I tried my hardest when I was doing AD IT UP," "I think AD IT UP would be helpful to other kids my age," "I would recommend AD IT UP to a friend," and "I agree with AD IT UP's message." An answer of "Strongly Agree" or "Agree" on these items indicates high and moderate acceptability, respectively. Each of these items will be assessed individually, not as an overall scale.
  Open-ended items will ask: what the student would change about AD IT UP, what the student liked about AD IT UP, what made AD IT UP fun, and what made AD IT UP not fun.

SECONDARY OUTCOMES:
Changes in intention to use tobacco products | baseline vs. 12 months
  Items adapted from the National Youth Tobacco Survey will be included in all 4 surveys. These items include the following with a 4-item response scale ranging from Definitely No to Definitely Yes:
  Do you think you will smoke a cigarette in the next month? Do you think you will smoke a cigarette at any time during the next year? If one of your best friends offered you a cigarette, would you smoke it?
  These items will be repeated for hookah, e-cigarettes, and cigars and cigarillos.
  Answering anything other than "Definitely No" on any item is considered "positive intention to use tobacco products." For example, if a student answers "Definitely Yes" to one cigarette item but "Probably No" to the other items, that student has positive intention to use cigarettes.
Changes in attitudes toward tobacco products | baseline vs. 12 months
  Items to measure attitudes toward tobacco products will be included in all 4 surveys. These items include the following with a 10-item response scale ranging from Strongly Disagree to Strongly Agree.
  E-cigarettes are not as bad for your health as other products. Using tobacco products at parties is fun. Tobacco products help you deal with problems or stress. Smoking helps people stay thin. People who use e-cigarettes are more fun to be around than people who don't use e-cigarettes.
  If someone starts using tobacco products every day, it is very hard for them to stop (reverse coded).
  Smoking makes a person look more attractive. It would be very easy for me to get e-cigarettes if I wanted them.
  Change in attitudes will be determined by the average increase or decrease in agreement with these items. These items will be assessed individually and as an overall scale (range 0-80, with higher scores indicating a worse outcome).
Changes in normative beliefs about tobacco products | baseline vs. 12 months
  Items to measure normative beliefs about tobacco products will be included in all 4 surveys. These items ask participants their rate how acceptable the following statements are among their friends using a 10-item response scale ranging from Very Acceptable to Very Unacceptable:
  It is OK for people your age to smoke cigarettes. It is OK for people your age to use e-cigarettes. It is OK for people your age to use hookahs. It is OK for people your age to smoke cigars or cigarillos. A wealthy person is more likely to use tobacco products than a poor person. A successful person is more likely to use tobacco products than an unsuccessful person.
  Changes in normative beliefs will be determined by the average increase or decrease in perceived acceptability of these statements. These items will be assessed individually, as well as an overall scale (range 0-60 with higher scores indicating a worse outcome).
Change in tobacco-related media literacy | baseline vs. 12 months
  Items to measure tobacco-related media literacy will be adapted from the Smoking Media Literacy Scale and included in all 4 surveys. The response scale for these 8 items is a 10-item scale from "Strongly Disagree" to "Strongly Agree."
  Changes in media literacy will be determined by the average increase or decrease in agreement with these items. These items will be assessed individually, as well as an overall scale (range 0-80, with higher scores indicating a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Sidani, PhD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Appropriate data from this project will be made available via the Open ScienceFramework, which is recommended by the University of Pittsburgh Library System.
  Shareable data generated during the project will include longitudinal survey results, which will contain both quantitative and qualitative information. Survey data will be sufficiently de-identified and formatted in a broadly accessible spreadsheet format. Generic participant ID numbers will be available to link data across survey timepoints. These data will be made available with accompanying metadata (i.e., file descriptors and codebook). For example, available codebooks will include labels and descriptors for each quantitative survey variable as well as definitions used for qualitative coding.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available approximately December 2023 and remain available for 3 years in accordance with the NIH Grants Policy Statement on Data Sharing.
Access Criteria: Interested researchers will contact the PI to request access.